CLINICAL TRIAL: NCT04457882
Title: Evaluation of the Safety of Intraperitoneal Laparoscopic Radical Prostatectomy With or Without Drainage Tube: a Singlecentre, Randomised Controlled, and Non-inferiority Study
Brief Title: Evaluation of the Safety of Intraperitoneal Laparoscopic Radical Prostatectomy With or Without Drainage Tube
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PD2020-001
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Laparoscopic Radical Prostatectomy; Intraperitoneal; Drainage Tube
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without Drainage Tube (Experimental): No place the drainage tube after the intraperitoneal laparoscopic radical prostatectomy
  Interventions: Behavioral: Intraperitoneal Laparoscopic Radical Prostatectomy Without Drainage Tube
- With Drainage Tube (Active Comparator): Place the drainage tube after the intraperitoneal laparoscopic radical prostatectomy
  Interventions: Behavioral: Intraperitoneal Laparoscopic Radical Prostatectomy With Drainage Tube

INTERVENTIONS:
Behavioral: Intraperitoneal Laparoscopic Radical Prostatectomy Without Drainage Tube — No place the drainage tube after the intraperitoneal Laparoscopic Radical Prostatectomy
  Arms: Without Drainage Tube
Behavioral: Intraperitoneal Laparoscopic Radical Prostatectomy With Drainage Tube — Place the drainage tube after the intraperitoneal Laparoscopic Radical Prostatectomy
  Arms: With Drainage Tube

SUMMARY:
This is a randomized controlled and non-inferiority trial in comparison of intraperitoneal laparoscopic radical prostatectomy without drainage tube between intraperitoneal laparoscopic radical prostatectomy with drainage tube in the safety in men with a localized prostate cancer.

DETAILED DESCRIPTION:
This trial is a prospective, single-centre, randomized controlled, and non-inferiority study in which all men with localized prostate cancer. This study aims to determine whether intraperitoneal laparoscopic radical prostatectomy without drainage tube is non-inferior to intraperitoneal laparoscopic radical prostatectomy with drainage tube in the safety in men with a localized prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. age: more than 18 years old, less than 85 years old;
2. Patient who pathologically diagnosed with prostate cancer and plan to undergo radical laparoscopic surgery for prostate cancer;
3. fully understand the clinical trial protocol and sign the informed consent;

Exclusion Criteria:

1. patients with surgical contraindications who cannot accept surgery;
2. patients with non-laparoscopic radical resection of prostate cancer;
3. patients with previous pelvic radiation therapy and complicated abdominal surgery;
4. patients judged by the investigator to be unsuitable to participate in the clinical trial;

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
The rate of adverse event | 3 month
  Any adverse event according to the Clavien-Dindo classification will be recorded

SECONDARY OUTCOMES:
Hemoglobin | 3 Months
  The difference between postoperative hemoglobin and preoperative hemoglobin
Physical recovery | 3 Months
  The time between the patient's first time out of bed and the end of the surgical procedure
Intestinal function recovery | 3 Months
  The first time to eat after the operation, the first time to exit gas after the operation,the first time to defecation after the operation
Abdominal effusion and cyst | 3 Months
  The ultrasound and CT to detect if there is abdominal effusion and cyst

CONTACTS AND LOCATIONS:
Overall Officials: Haifeng Wang, Principal Investigator — Shanghai East Hospital,Tongji University School of Medicine
Locations (1):
- Shanghai East Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality, China